CLINICAL TRIAL: NCT05570071
Title: A Randomized Controlled Clinical Study of the Use of Vaginal Radiofrequency Therapy in Treatment of Stress Urinary Incontinence.
Brief Title: A Study of the Use of Vaginal Radiofrequency Therapy in Treatment of SUI.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Li Yan, pfofessor, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022001
Record Dates: First submitted 2022-09-26; First posted 2022-10-06 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Urinary Incontinence, Stress
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vaginal radiofrequency (Experimental): vaginal radiofrequency therapy 4 times
  Interventions: Device: physical therapy
- electromyography biofeedback (Active Comparator): electromyography combined with biofeedback therapy 15 times
  Interventions: Device: physical therapy

INTERVENTIONS:
Device: physical therapy — medical treatment of pelvic floor

SUMMARY:
To investigate the immediate, short-term and long-term efficacy of vaginal radiofrequency therapy in the treatment of stress urinary incontinence, and to compare the efficacy of pelvic floor electromyography combined with biofeedback therapy in stress urinary incontinence.

DETAILED DESCRIPTION:
Before treatment, patients with mild and moderate stress urinary incontinence were diagnosed according to the diagnostic criteria through medical history inquiry and gynecological physical examination, and patients were screened according to the inclusion and exclusion criteria. After informing two treatment plans and signing the informed consent, they were randomly divided into vaginal radiofrequency therapy group and electrical stimulation combined biofeedback group. After being included in the test, one hour urine pad test was conducted, and IIQ-7, PISQ-12 and FSFI questionnaires were completed. IIQ-7, PISQ-12 and FSFI questionnaires were followed up 1, 3, 6 and 12 months after treatment. After 3 months and 1 year of treatment, 1 hour urine pad test was given again.

ELIGIBILITY:
Inclusion Criteria:

18-75 years old women with a sexual history, and patients with mild to moderate stress urinary incontinence.

Exclusion Criteria:

Severe cardiopulmonary insufficiency, acute pelvic inflammatory disease or other infectious stage, non-steroidal anti-inflammatory drugs and steroid hormones affecting collagen production factors, POP-Q-2 and above prolapse.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-20 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Urine leakage in 1-hour pad test | before therapy
  measure the urine leakage in 1-hour pad test
Change from urine leakage at 3 months | 3months after therapy
  measure the urine leakage in 1-hour pad test at 3 months
Change from urine leakage at 12 months | 12months after therapy
  measure the urine leakage in 1-hour pad test at 12 months

SECONDARY OUTCOMES:
incontinence impact questionnaire short form,IIQ-7 | before therapy
  Urinary incontinence may affect daily activities, interpersonal relationships or personal emotions.The minimum value is 0,and the maximum value is 21. Higher scores mean a worse outcome.
incontinence impact questionnaire short form,IIQ-7 | 3months after therapy
  Urinary incontinence may affect daily activities, interpersonal relationships or personal emotions.The minimum value is 0,and the maximum value is 21. Higher scores mean a worse outcome.
incontinence impact questionnaire short form,IIQ-7 | 12months after therapy
  Urinary incontinence may affect daily activities, interpersonal relationships or personal emotions.The minimum value is 0,and the maximum value is 21. Higher scores mean a worse outcome.
pelvic organ prolapsed-incontinence sexual questionnaire, PISQ-12 | before therapy
  The sexual desire，orgasm，pain，urine leakage in sex of the participants.The minimum value is 0,and the maximum value is 48.Higher scores mean a better outcome.
pelvic organ prolapsed-incontinence sexual questionnaire, PISQ-12 | 3months after therapy
  The sexual desire，orgasm，pain，urine leakage in sex of the participants.The minimum value is 0,and the maximum value is 48.Higher scores mean a better outcome.
pelvic organ prolapsed-incontinence sexual questionnaire, PISQ-12 | 12months after therapy
  The sexual desire，orgasm，pain，urine leakage in sex of the participants.The minimum value is 0,and the maximum value is 48.Higher scores mean a better outcome.
Female Sexual index，FSFI | before therapy
  Sex frequency，sexual satisfaction, physiological factors, affective factor , sexual partner factor. The minimum value is 0,and the maximum value is 124.Higher scores mean a better outcome.
Female Sexual index，FSFI | 3months after therapy
  Sex frequency，sexual satisfaction, physiological factors, affective factor , sexual partner factor. The minimum value is 0,and the maximum value is 124.Higher scores mean a better outcome.
Female Sexual index，FSFI | 12months after therapy
  Sex frequency，sexual satisfaction, physiological factors, affective factor , sexual partner factor.The minimum value is 0,and the maximum value is 124. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Li Yan, Study Director — Shandong First Medical University; Miao Yuan, Principal Investigator — Shandong First Medical University; Fangfang Zhao, Principal Investigator — Shandong First Medical University; Guangli Liu, Principal Investigator — Shandong First Medical University; Jing Li, Principal Investigator — Shandong First Medical University; Min Lu, Principal Investigator — Shandong First Medical University; Hongyan Niu, Principal Investigator — Shandong First Medical University; Dongyue Wang, Principal Investigator — Shandong First Medical University

IPD SHARING:
Plan to Share IPD: No